CLINICAL TRIAL: NCT06839508
Title: Comprehensive Management of Rectal Cancer
Acronym: CMRC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0073_CHIRURGIE
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Particular Case of Patients with Complete Response After CRT Traditionally, for patients with mid o: An initial opportunistic approach, also called Watch and Wait (W&W), involves monitoring patients who are considered to have a complete response after CRT or total neoadjuvant treatment, regardless of the initial stage. This approach was developed by Habr-Gama et al.
  Interventions: Other: Radio chemotherapy

INTERVENTIONS:
Other: Radio chemotherapy — The task involves identifying similarities in biopsy samples (prior to radio-chemotherapy treatment) to predict a hypothetical complete response.

SUMMARY:
study on the strategy we have adopted for rectal cancer treated with chemoradiotherapy in the case of a complete reponse ( surveillance vs. surgery) Particular Case of Patients with Complete Response After CRT. Traditionally, for patients with mid or lower rectal cancer, a protocol involving chemoradiotherapy followed by surgery 8 to 10 weeks after the end of radiotherapy and chemotherapy is systematically indicated after a post-chemoradiotherapy reassessment using pelvic MRI.

In a certain number of patients (25%), it was noted that the reevaluation through pelvic MRI after chemoradiotherapy shows complete tumor disappearance.

However, these patients were still operated on according to the standard procedure, and pathologists found no tumor in the surgical specimen (sterile specimen).

These are patients with a complete radiological and pathological response. In such cases, it is possible to resect the scar that remains at the site of the tumor (radiotherapy sequelae) and closely monitor the patient to detect recurrence in the short and medium term, thus avoiding mutilating surgery that impacts quality of life (fecal and gas incontinence, increased bowel movements, urinary and gynecological sexual disorders). This is known as the "Watch and Wait" strategy.

"Watch and Wait" Strategy. An initial opportunistic approach, also called Watch and Wait (W&W), involves monitoring patients who are considered to have a complete response after CRT or total neoadjuvant treatment, regardless of the initial stage. This approach was developed by Habr-Gama et al. in Brazil and published in 18 different articles, involving a cohort of 361 patients, with complete response rates ranging from 20% to 30%. Local recurrence rates varied from 5% to 25% depending on the articles and the timing of complete clinical response evaluation, while maintaining a 5-year disease-free survival rate of 52% and an overall survival rate of 85%. These series primarily included cT2 or cT3 tumors, but also cT4 tumors. Complete clinical response was defined as the absence of any clinical tumor residue (no tumor, no ulcer, and negative biopsy), and patients were monitored monthly.

However, the evaluation timeline for complete response varied across the articles, ranging from 8 weeks to 14 months.

At present, no official recommendations validate this strategy; it remains an expert opinion. The aim is to demonstrate that we could avoid surgery in patients with a complete response (we have favored rectal surgery for the majority of our patients due to organizational obstacles, patient-related issues, and the difficulty in applying rigorous surveillance in certain cases).

The purpose of this research is to improve our practices in managing rectal cancer in patients with a complete response.

ELIGIBILITY:
Inclusion Criteria:

* All patients managed in our facility who achieved a complete response after preoperative radio-chemotherapy.

Exclusion Criteria:

* Minor patients
* Non-responding patients, or partial responders.
* Anal canal cancer

Ages: 37 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
results heterogeneous. | 10/05/2024
  In all patients, a reevaluation was performed using a digital rectal exam (DRE), a rectosigmoidoscopy, a pelvic MRI, and a PET scan.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Saint Denis, Saint-Denis, France

REFERENCES:
- See also: site web — https://pubmed.ncbi.nlm.nih.gov/36972213